CLINICAL TRIAL: NCT02394249
Title: SIT LESS 3: The Effect of Low Intensity Physical Activity on Insulin Sensitivity, Mood and Cognitive Performance
Acronym: SIT LESS 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 143046; NL50688.068.14 (Registry Identifier: Medical Ethical Committee Maastricht University Hospital / University of Maastricht)
Record Dates: First submitted 2015-02-19; First posted 2015-03-20 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Overweight; Obesity
Keywords: Insulin Resistance; Cognition; Affect; Insulin; Lipids
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitting regime (Experimental): The subjects will follow the sitting regime during four days. Each day: 14 hours sitting, 1 hour walking and 1 hour standing and 8 hours sleeping.
  Interventions: Behavioral: Physical activity regime
- Sit Less regime (Experimental): Subjects will follow the sit less regime during four days. Each day will consist of 9 hours sitting, 4 hours walking, 3 hours standing and 8 hours sleeping. The walking and standing will be done in a minimum of eight bouts with a time interval of >1 hour. The subjects will be instructed to walk on a slow pace, i.e. 2-3 km/h, which is comparable to walking during shopping, walking to the office etc.
  Interventions: Behavioral: Physical activity regime

INTERVENTIONS:
Behavioral: Physical activity regime — Information already included in arm descriptions

SUMMARY:
Background of the study:

A sedentary lifestyle and obesity are well known risk factors of type 2 diabetes. The major focus of current guidelines for type 2 diabetes prevention is on energy balance. Physical activity guidelines recommend at least 30 minutes/day of moderate to vigorous physical activity (MVPA). However, no advice is given how the other 23.5 hours of the day should be spent. Several recent epidemiologic studies suggest that excessive sitting, independent of moderate to vigorous physical activity, has detrimental health effects. Another possibility to sit less is by increasing low intensity physical activities as slowly walking and standing. A recent published study of Duvivier and colleagues suggests that sitting less and replacing it by slowly walking and standing has a better effect on insulin action and cardiovascular risk factors than the combination of one hour MVPA per day and sitting the rest of the day in healthy subjects (Duvivier et al. PLOS ONE 2013). Until now this research is not performed in subjects with overweight/obesity.

Objective of the study:

To assess the effect of low intensity physical activity on plasma insulin levels, cognition and mood in subjects with overweight/obesity

Study population:

21 subjects between 40-80 years old with overweight/obesity

Intervention:

2 activity regimes of 4 days: a sitting regime and a "sit less" regime

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men and postmenopausal women: 40-80 years old
* BMI: 25.0 - 35.0 kg/m2
* Maximum 2.5 hours of MVPA per week (during last 3 months)
* Having a general practitioner
* Agreeing to be informed about medically relevant personal test-results by a physician
* Accessible veins on arms as determined by examination at screening

Exclusion Criteria:

* Reported participation in another biomedical trial which may have an effect on insulin sensitivity one month before the pre-study examination or during the study
* Blood donation in the past three months
* Reported participation in night shift work 2 weeks prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM.
* Consumption of >14 (women) or > 21 (men) alcoholic units per week
* Reported dietary habits: medically prescribed diet, slimming diet;
* Reported weight loss (>2kg) in the last three months prior to the screening;
* Not being able to execute at least three (out of four) cognition tests in the training session
* Not being able to execute the sit less try-out day
* Being an employee of Unilever or the collaborating research departments in Maastricht University Medical Centre
* Experimental drug use (during the last 3 months)
* Use of insulin, oral blood glucose lowering medication (metformin and/or SU-derivatives and/or DPP-IV inhibitors), corticosteroids or vitamin K antagonists in the last 3 months
* Fasting plasma glucose level > 6.9 mmol/L
* Medical conditions which make participation in the study not responsible which will be decided by a medical doctor during screening
* Other clinically relevant abnormalities in clinical chemistry at screening (to be judged by a medical doctor)
* Mental or physical disability which interferes with physical activity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Plasma insulin levels (measured as area under the curve during an oral glucose tolerance test) | one day after each regime
  To assess the effect of low intensity physical activity (LIPA) on plasma insulin levels (as measured as area under the curve during an oral glucose tolerance test)

SECONDARY OUTCOMES:
Insulin sensitivity (measured as Matsuda combined insulin sensitivity index during an oral glucose tolerance test) | one day after each regime
  To assess the effect of LIPA on insulin sensitivity
Plasma C-peptide | one day after each regime
  To assess the effect of LIPA on plasma C-peptide
Plasma glucose levels | one day after each regime
  To assess the effect of LIPA on plasma glucose levels
Plasma triglycerides | one day after each regime
  To assess the effect of LIPA on plasma triglycerides
Plasma total cholesterol | one day after each regime
  To assess the effect of LIPA on plasma total cholesterol
Plasma non-HDL cholesterol | one day after each regime
  To assess the effect of LIPA on plasma non-HDL cholesterol
Plasma HDL cholesterol | one day after each regime
  To assess the effect of LIPA on plasma HDL cholesterol
Plasma LDL cholesterol | one day after each regime
  To assess the effect of LIPA on plasma LDL cholesterol
Plasma free fatty acids | one day after each regime
  To assess the effect of LIPA on plasma free fatty acids
Plasma apolipoprotein B | one day after each regime
  To assess the effect of LIPA on plasma apolipoprotein B
Plasma apolipoprotein A | one day after each regime
  To assess the effect of LIPA on plasma apolipoprotein A
Mood (measured by the Affect Grid mood scale) | 2 days: last day of each regime and one day after each regime
  To assess the effect of LIPA on mood
Attention (measured by the Attention Network Task) | one day after each regime before and after the oral glucose tolerance test
  To assess the effect of LIPA on attention
Executive Function (measured by the Trail Making Test) | one day after each regime before and after the oral glucose tolerance test
  To assess the effect of LIPA on executive function
Memory (measured by the Rey Auditory Verbal Learning Task) | one day after each regime before and after the oral glucose tolerance test
  To assess the effect of LIPA on memory
Quality of life (measured by the Gill 32-item questionnaire) | last day of each regime
  To assess the effect of LIPA on quality of life
Sleep (measured by the 10-item Pittsburgh Sleep Quality Index) | last day of each regime
  To assess the effect of LIPA on sleep
Plasma C-reactive protein | one day after each regime
  To assess the effect of LIPA on plasma C-reactive protein
Plasma interleukin 1 | one day after each regime
  To assess the effect of LIPA on plasma interleukin 1
Plasma interleukin 6 | one day after each regime
  To assess the effect of LIPA on plasma interleukin 6
Plasma TNF-alpha | one day after each regime
  To assess the effect of LIPA on plasma TNF-alpha
Plasma interferon gamma | one day after each regime
  To assess the effect of LIPA on plasma interferon gamma
Plasma ICAM-1 | one day after each regime
  To assess the effect of LIPA on plasma ICAM-1
Plasma VCAM | one day after each regime
  To assess the effect of LIPA on plasma VCAM
Plasma serum amyloid A (SAA) | one day after each regime
  To assess the effect of LIPA on plasma SAA
Plasma E-selectine | one day after each regime
  To assess the effect of LIPA on plasma E-selectine
Plasma von Willebrand factor (vWF) | one day after each regime
  To assess the effect of LIPA on plasma vWF
Plasma PAI-1 | one day after each regime
  To assess the effect of LIPA on plasma PAI-1
To explore the association between plasma glucose, plasma insulin, insulin sensitivity and mood, cognitive performance, quality of life and sleep | one day after each regime
Blood pressure | one day after each regime
Heart rate | one day after each regime

CONTACTS AND LOCATIONS:
Overall Officials: Hans H Savelberg, PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Human Movement Science, Maastricht University, Maastricht, Maastricht, Netherlands

REFERENCES:
- [Background] Duvivier BM, Schaper NC, Bremers MA, van Crombrugge G, Menheere PP, Kars M, Savelberg HH. Minimal intensity physical activity (standing and walking) of longer duration improves insulin action and plasma lipids more than shorter periods of moderate to vigorous exercise (cycling) in sedentary subjects when energy expenditure is comparable. PLoS One. 2013;8(2):e55542. doi: 10.1371/journal.pone.0055542. Epub 2013 Feb 13. PMID 23418444
- See also: Related Info — http://www.plosone.org/article/metrics/info%3Adoi%2F10.1371%2Fjournal.pone.0055542